CLINICAL TRIAL: NCT07056023
Title: Multicenter Trial on Surgical Outcome and Quality of Life in Juxta-medullary Tumors
Acronym: EURJMT
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Technical University of Munich (Other); University Hospital Freiburg (Other); Medical University of Cologne (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Michael Schwake, Director of the Neurosurgery Spine Section, University Hospital Muenster
Other Study IDs: EURJMT
Record Dates: First submitted 2025-05-19; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Intraspinal Tumor; Juxtamedullary Tumor
Keywords: intra-dural tumors; spinal meningioma; spinal schwannoma; spinal ependymoma
MeSH Terms: conditions — Spinal Cord Neoplasms; Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objectives: Primary objectives are to assess and define benchmarks of the surgical outcome in the form of extent of resection, functionality, and quality of life after resection of juxta medullary tumors Secondary objectives: Assessment of variables leading to better outcome through regression analysis: 1. Influence of surgical approach on functionality, pain, and quality of life 2. Comparison between patient with severe neurological (McCormick scale 3-5) to patients with mild deficits (McCormick scale 1-2) 3. Role of intraoperative monitoring (IOM) in extent of resection and neurological deficits Assessment of treatment variations: 1. Assessment of risk factors for incomplete resection 2. Non inferiority of unilateral approach to achieve gross total resection of spinal meningioma, schwannoma and cauda ependymoma 3. Role of bed rest after surgery to prevent cerebro-spinal fluid leakage 4. Influence of laminectomy on cerebro-spinal fluid leakage Quality indicators: assessments of length of hospital stay, 30- and 90-days re-admissions, 30- and 90-days re-surgery, nosocomial infections

DETAILED DESCRIPTION:
Introduction

1. Background information Juxta-medullary tumors are mostly benign tumors in the spinal canal that may cause neurological deficits due to spinal cord or nerve root compression. The knowledge about the natural course of the disease, optimal treatment regarding timing of surgery and surgical approach are based on case series from different institutions around the world. Moreover, little is known about the long-term clinical and functional outcome after tumor resection, indicators of quality of treatment and quality of life after surgery.

Main treatment option of juxta-medullary tumors is a neurosurgical resection. The main goal of the surgery is to decompress the neuro structures in order to reveal neurological deficits. However, achieving gross total resection (GTR) is important in order to achieve long progression free survival (PFS).

Therefore, the surgeon should choose the appropriate surgical approach to achieve these goals. Several publications show that GTR, whenever possible, is essential, as subtotal resection is the main reason of tumor regrowth or recurrence. Moreover, revision surgery due to tumor recurrence is one of the main risk factors of unfavorable outcome, probably to intradural adhesions, related to the first procedure. Due to the mostly benign nature of juxtamedullary tumors, it would be very difficult to evaluate overall survival (OS) and progression free survival (PFS) within this progressive registry in the short run. For this reason, data should be kept for late cohort analysis after longer intervals. Probably up to 20 years, as previous publications reported recurrence of spinal meningioma after GTR 10 years or more after surgery.

On the other hand, too large exposure may lead to impaired recovery after surgery, eventual higher blood loss during surgery and thus longer stay in hospital (LOS) and impaired quality of life. Moreover, extensive bone resection may lead to spinal instability requiring instrumentation, during index surgery or during further follow up in case of postoperative deformity).

In addition to the oncological outcome, the neurological outcome is also very important. Depending on the localization of the tumor, its form and compression of intra-spinal structures such as the spinal cord or nerve roots many patients develop neurological deficits. Besides GTR the other goal of resection is the neurological recovery of these patients. Previous reports show that the time point of surgery is important in order to achieve full recovery. However, most of the data is derived from retrospective case series. One of the aims of this registry is to prove this hypothesis. These neurological deficits are, as mentioned above, related to the localization of the tumor within the spine, Tumors in the cervical spine would cause mainly gait ataxia, spasticity, and weakness in the upper extremities while tumors in the lumbar spine would lead to deficits in the lower extremities in combination to disturbances of bladder, bowl, and sexual functions. These functions should be evaluated and monitored, before and after treatment.

Other concerns are safety requirements in order to prevent peri-operative complications. For example, the role of intra-operative neurophysiological monitoring. Some authors recommend the utilization intra operative monitoring, however, the evidence level is very low. Other open questions are for example the utility of microscope, methods for dura closure and thrombosis prevention.

On the other hand, some tumors can be treated with irradiation, some studies showed efficacy of this method mainly in the case of Schwannomas and meningiomas. In case of residual tumor or tumor progression irradiation can be also performed to prevent further growth.

Lastly, in comparison to the methods mentioned above, a wait-and-see approach can be used for asymptomatic patients or those with mild symptoms. In this case, clinical and imaging examinations are performed at regular intervals to check the neurological status and the tumor. This can also be done for longer periods of time because of the benign nature of these tumors with the slow growth. in case of new neurological deficits of or progression surgical treatment should be advocated. Overall, it is not certain at what point therapy is indicated, especially in asymptomatic patients. Because many of these tumors are discovered by coincidence during imaging, which was performed due to other symptoms.

2 Rationale of the study The rationale of the trial is to define benchmarks on quality of life, functionality and neurological outcome after resection of juxtamedullary tumors. Furthermore, to assess and define benchmarks of quality indicators of the treatment. These measurements would be essential for future studies.

Further rationales are to find out the optimal timing, method, and approach to treat juxta-medullary tumors. Because of the low incidence of juxta-medullary tumors, a multi-center trial seems to be essential. This would allow us to analyze a large number of patients, much more than any other published paper. Moreover, the different protocols and standards approaches in each center would allow conducting Comparative Effectiveness Research (CER).

3 Aims The goal of this study is to establish a multicenter cohort of patients operated on juxtamedullary tumors. With especial emphasis on functional outcome, quality indicators (QI) and quality of life after surgery three months after surgery. Causes of unfavorable outcome should be determined.

The main hypothesis is that early and less-invasive surgery with maximal extents of resection would lead to a more favorable outcome. In the future the registry would help assessing further hypothesis can be answered on the base of comparative effectiveness research (CER), examples of these hypothesis are:

1. Functional and neurological outcome in comparison to preoperative status. Comparison between Panties with good preoperative McCormick score (1-2) and those with a high preoperative score (3-5).
2. Risk-factors for non-favorable outcome
3. Non-Inferiority to achieve gross total resection via unilateral approaches
4. Question whether laminectomy as approach may cause mor pain and impact quality of life
5. Risk factors for the development of CFS Leaks
6. Does bed rest prevent CSF leaks
7. Does laminectomy elevate the risk of CSF leaks
8. Does the utility of intraoperative neurophysiological monitoring (IOM) influence surgical outcome: rate of GTR and neurological outcome
9. Rate of postoperative kyphosis and deformity in laminectomy in comparison to non-laminectomy
10. Is facetectomy required for GTR of dumbbell tumors?
11. Risk factors for non-complete resection

Primary outcomes are determined by:

Quality of life based on the questionnaire (EQ-D5) Extent of tumor resection (see CRF): according to surgeon: 1. Meningioma: Simpson grade 1 and 2 2. Schwannoma: complete resection, including nerve root 3. Cauda ependymoma: complete resection, including filum terminale according to postoperative MRI, 3 months after surgery 4. Other: surgeon's decision Neurological status (McCormick Score) (see CRF), 3 months after surgery Secondary Outcome Imaging: preoperative and postoperative MRI Volumetry Spinal canal occupancy ratio in %

Further patient reported outcomes:

Functionality: Neck disability index (NDI) for tumors in the cervical spine, Oswestry disability index (ODI) for tumors in the thoracic and lumbar spine (see CRF) Local and radicular pain (VAS 1-10) (see CFR) Neurological status: motor function of each limb, ataxia and gait (mJOA score) (see CRF) HADS score- based score for anxiety Questionnaire on bladder, bowl, sexual functionality

Quality indicators (QI):

Length of hospital stay 30- and 90-days readmission Nosocomial infections Blood loss Duration of surgery Progression of the disease or recurrence Other adverse events Mortality Assessment of adverse events according to Common Terminology Criteria for Adveres Events (CTCAE) 5.0 and severity according to the Ibañez scale (see CRF) CSF leakage is defined as one, when CSF leakage is identified on imaging of clinicaly and treatment is required: operative or conservative (Lumbar drain for example) Postoperative kyphosis of deformity is defined, when symptomatic (for example pain) or evident on imaging (for example kyphotic fracture on MRI) Methodology All patients treated in one of the study centers are recorded in a databank (Redcap, see below), which includes information about admission, symptoms, other diseases, treatment, quality indicators and questionnaires regarding quality of life and functionality. Data should be recorded in an anonymized in each center (see below).

For the analysis the CRF includes information about admission, surgery, discharge, and 3 months (90 days) after surgery. In addition, patients should fill out questionnaires on quality of life (EQ-D5) and functionality (ODI or NDI). Later, yearly visits can be completed to have long term results in the future regarding progression free survival (PFS) and overall survival (OS). The CRF is attached to this document.

Univariate and multivariate statistics would be applied to prove which variables might lead to a favorable or unfavorable outcome.

A minimum number of one hundred (N=100) inclusions seems to be adequate in order to perform reasonable analysis. In the event of nonsufficient recruitment, results and further recruitment would be discussed two years after initiation of the study, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age ≥18 years, patients treated on intraspinal, extra medullary tumor
* Patients must have sufficient cognitive and language skills to give informed consent

Exclusion Criteria:

* Absence of informed consent
* Lack of ability to consent
* Primary bone tumors invading the intra-spinal space
* Vertebral metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, age ≥18 years, patients treated on intraspinal, extra medullary tumor
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life based on the questionnaire | prior and 3 months after resection
  The EuroQol 5-Dimension questionnaire (EQ-5D) is a standardized measure of health-related quality of life. It includes five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each rated on 3 or 5 levels, and a visual analogue scale (EQ VAS) from 0 (worst health imaginable) to 100 (best health imaginable). Higher EQ VAS scores indicate better health status. The descriptive system can also be converted to an index score ranging typically from <0 (worse than death) to 1 (perfect health), where higher values reflect better health.
Extent of tumor resection | 3 months after resection
  1. Meningioma: Simpson grade 1 and 2 2. Schwannoma: complete resection, including nerve root 3. Cauda ependymoma: complete resection, including filum terminale according to postoperative MRI, 3 months after surgery 4. Other: surgeon's decision
Neurological status | prior to surgery and 3 months after surgery
  The McCormick Functional Classification Scale for Spinal Cord Tumors assesses functional impairment in patients with intramedullary spinal tumors. It ranges from Grade I (minimal symptoms, fully active) to Grade IV (severe disability, dependent). The scale has four grades, with Grade I as the best and Grade IV as the worst outcome. Higher grades indicate greater neurological impairment and reduced functional independence.

SECONDARY OUTCOMES:
Tumor Volume | prior to surgery and 3 months after surgery
  The Tumor Volume on MRI Scans measures the three-dimensional size of a tumor using magnetic resonance imaging. It is typically calculated by multiplying tumor dimensions (length × width × height) and applying a correction factor (e.g., ×0.5 for ellipsoid shapes). Volume is expressed in cubic millimeters (mm³) or centimeters (cm³). There is no fixed minimum or maximum, as values depend on tumor size
Spinal Canal Ratio | prior surgery and 3 moths after surgery
  The Spinal Canal Ratio (also called the Spinal Canal Occupation Ratio) quantifies spinal canal narrowing, typically in cases of spinal stenosis or tumors. It is calculated as the ratio of the space occupied by the lesion (e.g., tumor or disc) to the total area of the spinal canal on axial imaging. Values range from 0 (no compression) to 1 (100% occupation of the canal). Higher values indicate worse outcomes, reflecting more severe canal compromise and potential cord compression.
Functionality: Oswestry disability index (ODI) for tumors in the thoracic and lumbar spine | prior and 3 months after surgery
  The Oswestry Disability Index (ODI) is a patient-reported questionnaire used to assess disability due to lower back pain. It includes 10 sections covering pain intensity and functional limitations (e.g., walking, lifting, sleeping), each scored from 0 to 5. The total score is converted to a percentage from 0% (no disability) to 100% (maximum disability). Higher scores indicate worse outcomes, reflecting greater functional impairment. The ODI is widely used to evaluate treatment effectiveness and monitor progress in patients with spinal disorders.
Funtionality: Neck disability index (NDI) for tumors in the cervical spine | prior surgry and 3 months after surgery
  The Neck Disability Index (NDI) is a validated, patient-reported questionnaire used to measure self-rated disability related to neck pain. It includes 10 items covering pain intensity and daily activities (e.g., personal care, lifting, concentration), each scored from 0 to 5. The total score ranges from 0 to 50, which is often expressed as a percentage (0% to 100%), where 0 indicates no disability and 100 indicates complete disability. Higher scores represent worse outcomes, reflecting greater functional impairment due to neck pain.
Local and radicular pain | prior and 3 months after surgery
  The Visual Analogue Scale (VAS) is a simple and widely used tool to measure subjective experiences such as pain intensity. Patients rate their pain on a continuous scale from 0 to 10 or 0 to 100, with 0 representing "no pain" and the maximum value (10 or 100) indicating the "worst pain imaginable." Higher scores reflect worse outcomes, corresponding to greater pain severity. The VAS is quick to administer and sensitive to changes over time, making it useful for monitoring treatment effects.
Neurological status | prior and 3 months after surgery
  Motor, sensory, ataxia, and gait disturbances are recorded as yes or no.
Motor deficits | prior surgery and 3 months after surgery
  The Medical Research Council (MRC) Scale for Muscle Strength is a standardized tool used to grade muscle power in patients with motor deficits. Each muscle group is scored from 0 to 5, where 0 indicates no muscle contraction and 5 indicates normal strength. The total score can range from 0 to 5 per muscle group, with higher scores indicating better outcomes and less motor impairment. The scale is widely used in neurology and rehabilitation to assess and monitor motor function over time.
anxiety and depression | prior and 3 months after surgery
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire used to screen for symptoms of anxiety and depression in medically ill patients. It consists of 14 items, split into two subscales: HADS-A (anxiety) and HADS-D (depression), each ranging from 0 to 21. Each item is scored from 0 to 3. The total HADS score ranges from 0 to 42, with higher scores indicating worse outcomes, i.e., greater psychological distress. Scores ≥8 on either subscale suggest clinically relevant symptoms. HADS does not assess motor deficits.
bladder functionality | prior and 3 months after surgery
  questionaire on functionality:
  Sensation in the "saddle" area (buttocks, medial hips)
  * Normal
  * Paresthesia
  * Reduced sensation
  * Absent sensation
  Bladder function:
  * Normal function
  * Mild dysfunction (occasional incontinence, but mostly continent)
  * Moderate dysfunction (frequent incontinence, but some control)
  * Severe dysfunction (total incontinence)
Bowl functionality | prior surgery and 3 months after surgery
  The Low Anterior Resection Syndrome (LARS) Score is a validated questionnaire used to assess bowel dysfunction after low anterior resection for rectal cancer. It includes 5 items covering incontinence, frequency, clustering, urgency, and gas control. Each response has a weighted score, with a total score ranging from 0 to 42. Scores are classified as No LARS (0-20), Minor LARS (21-29), or Major LARS (30-42). Higher scores indicate worse outcomes, reflecting more severe bowel dysfunction and impact on quality of life.
Sexual funtionality | prior and 3 months after surgery
  Questionaire:
  Males
  * Normal erectile and ejaculatory function
  * Mild erectile or ejaculatory dysfunction (able to have intercourse with mild difficulty)
  * Moderate erectile or ejaculatory dysfunction (intercourse possible with significant difficulty or partial erection)
  * Severe erectile or ejaculatory dysfunction (intercourse rarely or not possible)
  * Complete loss of erectile and ejaculatory function Females
  * Normal sexual function
  * Mild dysfunction (decreased arousal or lubrication, but able to have intercourse) Moderate dysfunction (significant difficulty with arousal or lubrication, painful intercourse)
  * Severe dysfunction (intercourse rarely or not possible due to dysfunction)
  * Complete loss of sexual function
Length of hospital stay | Perioperative/Periprocedural
  Length of hospital stay in days after asurgery. Day 0 is day of surgery
30-days readmission | 3 months after surgery
  Whether the patient was admitted to the hospital within 30 days after surgery
90-days readmission | 3 months after surgery
  Whether the patient was admitted to the hospital within 30 days after surgery
Nosocomial infections | Perioperative/Periprocedural and 3 motnhs after surgery
  Whether the patient had a nosocomial infection after surgery. A nosocomial infection, also known as a hospital-acquired infection (HAI), is an infection that develops 48 hours or more after hospital admission or within 30 days after receiving healthcare, which was not present or incubating at the time of admission. Common types include pneumonia, urinary tract infections, surgical site infections, and bloodstream infections. These infections often involve antibiotic-resistant organisms and can increase morbidity, mortality, and healthcare costs.
estbimated blood loss | Perioperative/Periprocedural
  The Estimated Blood Loss (EBL) During Surgery is a clinical measure used to approximate the volume of blood a patient loses during an operation. It is typically recorded in milliliters (mL), based on visual assessment, suction canister volume, and gauze saturation. There is no fixed minimum or maximum, but values can range from a few milliliters to several liters, depending on the procedure. Higher EBL values indicate worse outcomes, as they may reflect surgical complexity, increased risk of transfusion, and postoperative complications.
Duration of surgery | Perioperative/Periprocedural"
  Duration of surgery in minutes
Progression of the disease or recurrence | 3 months after surgery
  tumor growth visible on MRI
adverse events | 3 months after surgery
  adverse events not mentioned in the protocol should be also recored. The Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 is a standardized classification system developed by the U.S. National Cancer Institute to document and grade the severity of adverse events (AEs) in clinical trials. It includes over 800 terms covering organ systems, symptoms, and lab abnormalities. Each adverse event is graded from Grade 1 (mild) to Grade 5 (death related to AE). CTCAE ensures consistent reporting, supports safety monitoring, and facilitates comparison of safety profiles across studies.
Mortality | 3 months after surgery
  death of patients within 90 days after surgery
advers events _2 | Perioperative/Periprocedural and 3 months after surgery
  The Ibañez Scale is a classification system used to grade adverse events and complications following spinal surgery. It categorizes complications based on their severity and the need for intervention, helping to standardize outcome reporting. The scale ranges from Grade I (minor, requiring no treatment) to Grade IV (life-threatening or resulting in death). It allows clinicians to objectively assess and compare postoperative morbidity, supports clinical decision-making, and improves transparency in surgical outcome reporting.
CSF leakage | Perioperative/Periprocedural and 3 months after surgery
  CSF leakage is defined as one, when CSF leakage is identified on imaging of clinicaly and treatment is required: operative or conservative (Lumbar drain for example)
Postoperative kyphosis | 3 months after surgery
  Postoperative kyphosis of deformity is defined, when symptomatic (for example pain) or evident on imaging (for example kyphotic fracture on MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Muenster, Münster, Nordrhien Westfalen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT07056023/Prot_000.pdf